CLINICAL TRIAL: NCT05332405
Title: SPY Angiography To Determine the Extent of Nerve Release After Nerve Decompression
Brief Title: SPY Angiography To Assist With Ulnar Nerve Transposition at the Elbow
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Obsolete study
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-01449
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Cubital Tunnel Syndrome
MeSH Terms: conditions — Cubital Tunnel Syndrome | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Participants will have planned surgical procedure to repair the median or ulnar nerve compression. During the procedure, the doctor will administer a small injection of indocyanine green (ICG) and laser angiography using the SPY Elite device will be used to evaluate blood flow and extent of nerve decompression at the surgical site. Participation will also involve filling out two questionnaires on pain and function level and an examination of hand strength and range of motion.
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — The subject will receive 3mL of ICG followed by 10 mL of sterile saline intravenously as per the Spy Elite protocol. Within minutes of the injection, the SPY machine will be turned on and focused on the nerve. The SPY machine gives a digital read out of the % fluorescence when the dye reaches the nerve. This number correlates with blood flow or vascularity.
  Other Names: SPY AGENT GREEN

SUMMARY:
Patients with vascular disease, thyroid disease or an allergy to indocyanine green (ICG) will be excluded. Patients with either median or ulnar nerve compression will be treated with nerve decompression. SPY angiography will be used to assess the vascularity of the nerve both pre and post release as the primary outcome measure.

DETAILED DESCRIPTION:
The purpose of this study is to use laser imaging to determine the extent of nerve decompression (release) while patients are still in surgery. Commonly, this is determined by electrodiagnostic tests or physical examination. The researchers will use the SPY elite device along with an injection of a drug called SPY Agent green (indocyanine green) in an imaging procedure called fluorescence angiography to visualize the change in blood supply to the nerve, following the nerve decompression surgery and assess if SPY is a useful tool for evaluating the success of nerve decompression surgery. The use of fluorescence angiography with the SPY elite device and SPY agent green is Food and Drug Administration (FDA) approved.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older; male and female patients
* Ulnar Nerve Compression at the Elbow
* Failed conservative treatment (i.e. hand therapy, pain medications, splinting)
* Able to provide informed consent

Exclusion Criteria:

* Pregnancy/breastfeeding
* Thyroid Disease
* Vascular Disease
* Known allergy to any study drug

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in level of Fluorescence before and after nerve release. | 2 weeks, 6 weeks, 3 months, 6 months, and 12 months visits
  Assessed by comparing the SPY angiography value before and after nerve release surgery

SECONDARY OUTCOMES:
nerve function determined by grip strength | 2 weeks, 6 weeks, 3 months, 6 months, and 12 months visits
  Assessed by comparing the value of grip strength at each follow-up visits to the value of grip strength before nerve release surgery
Change in Monofilament sensory testing | 2 weeks, 6 weeks, 3 months, 6 months, and 12 months visits
  Assessed by comparing the Monofilament sensory testing score at each follow-up visit to the Monofilament sensory testing score before nerve release surgery
Change in DASH Score | 2 weeks, 6 weeks, 3 months, 6 months, and 12 months visits
  DASH score at each follow-up visit does not differ from that before nerve release surgery. Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale. A higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability. The score on the test ranges is from 0 (no disability) to 100 (most severe disability).

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Hacquebord, MD, Study Director — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be used for this study